CLINICAL TRIAL: NCT02289820
Title: A Phase 1b Study to Evaluate the Safety and Immunogenicity of MEDI7510 in Older Adults
Brief Title: A Study to Evaluate the Safety and Immunogenicity of MEDI7510 in Older Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: D4420C00004
Record Dates: First submitted 2014-11-10; First posted 2014-11-13 (Estimated); Results first posted 2018-02-19 (Actual); Last update posted 2018-03-15 (Actual); Status verified 2018-02

CONDITIONS: Respiratory Syncytial Virus (RSV)
Keywords: RSV; Older adults; MEDI7510; Vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- MEDI7510 (120 mcg sF + 1 mcg GLA), Cohort 1 (Experimental): Participants will receive a single dose of MEDI7510 (120 microgram [mcg] respiratory syncytial virus [RSV] soluble fusion protein [sF] plus 1.0 mcg glucopyranosyl lipid A in 2% volume per volume stable emulsion) administered by intramuscular (IM) injection on Day 1.
  Interventions: Biological: MEDI7510
- MEDI7510 (120 mcg sF + 2.5 mcg GLA), Cohort 2 (Experimental): Participants will receive a single dose of MEDI7510 (120 mcg RSV sF plus 2.5 mcg glucopyranosyl lipid A in 2% volume per volume stable emulsion) plus IIV or MEDI7510 plus placebo administered by IM injection in contralateral arms on Day 1.
  Interventions: Biological: MEDI7510; Biological: IIV
- MEDI7510 (120 mcg sF + 5 mcg GLA), Cohort 3 (Experimental): Participants will receive a single dose of MEDI7510 (120 mcg RSV sF plus 5.0 mcg glucopyranosyl lipid A in 2% volume per volume stable emulsion) plus IIV or MEDI7510 plus placebo administered by IM injection in contralateral arms on Day 1.
  Interventions: Biological: MEDI7510
- MEDI7510 (80 mcg sF + 2.5 mcg GLA), Cohort 4 (Experimental): Participants will receive a single dose of MEDI7510 (80 mcg RSV sF plus 2.5 mcg glucopyranosyl lipid A in 2% volume per volume stable emulsion) administered by IM injection on Day 1.
  Interventions: Biological: MEDI7510
- Inactivated Influenza Vaccine (IIV) (Active Comparator): Participants will receive a single dose of IIV by intramuscular injection in contralateral arms on Day 1.
  Interventions: Biological: IIV

INTERVENTIONS:
Biological: MEDI7510 — RSV sF antigen plus adjuvant
  Arms: MEDI7510 (120 mcg sF + 1 mcg GLA), Cohort 1; MEDI7510 (120 mcg sF + 2.5 mcg GLA), Cohort 2; MEDI7510 (120 mcg sF + 5 mcg GLA), Cohort 3; MEDI7510 (80 mcg sF + 2.5 mcg GLA), Cohort 4
Biological: IIV — Marketed Inactivated Influenza Vaccine
  Arms: Inactivated Influenza Vaccine (IIV); MEDI7510 (120 mcg sF + 2.5 mcg GLA), Cohort 2

SUMMARY:
The goal of this study is to evaluate the safety, tolerability and immunogenicity of ascending doses of adjuvant in combination with a single dosage level of RSV sF in adults 60 years or older who are healthy or who have stable, chronic underlying medical conditions. This study will also provide preliminary safety and immunogenicity data to support concurrent dosing of MEDI7510 with influenza vaccine (IIV), and to assess the safety of MEDI7510 at a dose previously assessed in the Phase 1a study.

DETAILED DESCRIPTION:
A Phase 1b, double-blind, randomized, controlled cohort escalation study evaluating the safety, tolerability and immunogenicity of MEDI7510.

Approximately 264 subjects will be enrolled at approximately 5 study centers in the US and randomized by cohort (Cohort 1 [4:1]; Cohorts 2 and 3 [8:8:3]; Cohort 4 [5:1]) to receive a single intramuscular dose of 1 study vaccine (Cohorts 1 and 4) or a single intramuscular dose of each of 2 study vaccines (Cohorts 2 and 3) administered in contralateral arms.

Cohort 1: MEDI7510 formulation (n = 40) or IIV (n = 10) Cohort 2: MEDI7510 formulation and placebo (n = 40) or MEDI7510 formulation and IIV (n = 40) or placebo and IIV (n = 15) Cohort 3: MEDI7510 formulation and placebo (n = 40) or MEDI7510 formulation and IIV (n = 40) or placebo and IIV (n = 15) Cohort 4: MEDI7510 formulation (n = 20) or IIV (n = 4)

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 60 years
* Ambulatory or ambulatory with assistance (not institutionalized, bedridden, or homebound)
* Weight greater than 90 lbs
* Hemoglobin greater than or equal to 10.5 g/dL for women and greater than or equal to 11 g/dL for men
* Subject able to complete follow-up period of 360 days after dosing

Exclusion Criteria:

* History of allergy to: any component of the vaccine; IIV or intolerance of IIV; eggs in adulthood
* Receipt of seasonal flu shot within 60 days prior to dosing
* Any unstable acute or chronic medical condition, including one that has resulted in change in therapy (medication or other) in the 30 days prior to randomization or hospitalization in the previous year or might be predicted to result in hospitalization in the year after enrollment. Subjects with severe, untreated or uncontrolled underlying medical disease that might either compromise subject safety or affect the ability to assess safety of the investigational product are excluded. Medications taken on an as-needed basis are permitted to start or stop during the 30 days prior to randomization unless they are medications not previously taken by the subject
* Clinically significant abnormalities in screening laboratory assessments or screening ECG
* History of hepatitis B or hepatitis C infection
* History of Guillain-Barré syndrome
* Cognitive disorder such that informed consent cannot be obtained directly from the subject
* Previous vaccination against RSV
* History of or current autoimmune disorder
* Immunosuppression caused by disease, including human immunodeficiency virus (HIV) infection, or medications. Any oral prednisone dosing within 30 days of enrollment or planned dosing within the 360-day follow-up period would disqualify. Expected need for immunosuppressive medications during the 360-day follow-up period would disqualify
* History of splenectomy or of condition affecting splenic function (eg, hemoglobinopathy)
* History of cancer within preceding 5 years other than treated non-melanoma skin cancer
* Body Mass Index 40 or higher
* Receipt of any nonstudy vaccine within 30 days prior to study dosing or expected receipt of nonstudy vaccine within 30 days after study dosing
* Receipt of any investigational product in the 90 days prior to randomization or expected receipt of investigational product during the period of study follow-up
* Receipt of immunoglobulins or blood products within 4 months of study dosing (120 days) or expected receipt of investigational product during the period of study follow-up
* Current bleeding or clotting disorder including use of anticoagulants other than drugs with anti-platelet activity (such as nonsteroidal anti-inflammatory drugs, clopidogrel, ticagrelor or aspirin)
* Expected receipt of antipyretic or analgesic medication on a daily or every other day basis from randomization through 72 hours after receipt of IP (Note: A daily dose of aspirin is not considered a contraindication to enrollment.)
* Subjects who have significant scarring, tattoos, abrasions, cuts, or infections over the deltoid region of both arms that, in the investigators opinion, could interfere with evaluation of injection site local reactions
* Concurrent enrollment in another clinical study that involves any invasive clinical procedure, including phlebotomy
* History of alcohol or drug abuse or psychiatric disorder that, in the investigators opinion, would affect the subject's safety or compliance with study
* Employees of individuals directly involved with the conduct of the study, individuals who themselves are involved with the conduct of the study, or immediate family members of such individuals

Ages: 60 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 363 (Actual)
Dates: Start 2015-01-05 (Actual); Primary Completion 2016-02-24 (Actual); Study Completion 2016-02-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith Falloon, MD, Study Director — MedImmune LLC; Eric Sheldon, MD, Principal Investigator — Miami Research Associates; Craig Curtis, MD, Principal Investigator — Compass Research; John Ervin, MD, Principal Investigator — The Center for Pharmaceutical Research; Wayne Harper, MD, Principal Investigator — Wake Research Associates; H. Keipp Talbot, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (5):
- United States (5):
  - Research Site, Orlando, Florida
  - Research Site, South Miami, Florida
  - Research Site, Kansas City, Missouri
  - Research Site, Raleigh, North Carolina
  - Research Site, Nashville, Tennessee

REFERENCES:
- [Derived] Chang LA, Phung E, Crank MC, Morabito KM, Villafana T, Dubovsky F, Falloon J, Esser MT, Lin BC, Chen GL, Graham BS, Ruckwardt TJ. A prefusion-stabilized RSV F subunit vaccine elicits B cell responses with greater breadth and potency than a postfusion F vaccine. Sci Transl Med. 2022 Dec 21;14(676):eade0424. doi: 10.1126/scitranslmed.ade0424. Epub 2022 Dec 21. PMID 36542692
- [Derived] Falloon J, Talbot HK, Curtis C, Ervin J, Krieger D, Dubovsky F, Takas T, Yu J, Yu L, Lambert SL, Villafana T, Esser MT. Dose Selection for an Adjuvanted Respiratory Syncytial Virus F Protein Vaccine for Older Adults Based on Humoral and Cellular Immune Responses. Clin Vaccine Immunol. 2017 Sep 5;24(9):e00157-17. doi: 10.1128/CVI.00157-17. Print 2017 Sep. PMID 28679495

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 363 participants were screened. Of these, 264 participants were enrolled.
Pre-assignment Details: A total of 264 participants were enrolled in the study. Of the 264 randomized participants, 3 participants did not receive the study drug. 261 participants were included in the As-treated Population.
Groups:
- MEDI7510 (120 mcg sF + 1 mcg GLA), Cohort 1: Participants received single dose of MEDI7510 (120 microgram [mcg] respiratory syncytial virus [RSV] soluble fusion protein [sF] plus 1.0 mcg glucopyranosyl lipid A in 2% volume per volume stable emulsion) administered by intramuscular (IM) injection on Day 1.
- MEDI7510 (80 mcg sF + 2.5 mcg GLA), Cohort 4: Participants received single dose of MEDI7510 (80 mcg RSV sF plus 2.5 mcg glucopyranosyl lipid A in 2% volume per volume stable emulsion) administered by IM injection on Day 1.
- Inactivated Influenza Vaccine (IIV): Participants received single dose of IIV by intramuscular injection in contralateral arms on Day 1.
- MEDI7510 (120 mcg sF + 2.5 mcg GLA) + Placebo, Cohort 2: Participants received single dose of MEDI7510 (120 mcg RSV sF plus 2.5 mcg glucopyranosyl lipid A in 2% volume per volume stable emulsion) plus placebo administered by IM injection in contralateral arms on Day 1.
- MEDI7510 (120 mcg sF + 2.5 mcg GLA) + IIV, Cohort 2: Participants received single dose of MEDI7510 (120 mcg RSV sF plus 2.5 mcg glucopyranosyl lipid A in 2% volume per volume stable emulsion) plus IIV administered by IM injection in contralateral arms on Day 1.
- MEDI7510 (120 mcg sF + 5 mcg GLA) + Placebo, Cohort 3: Participants received single dose of MEDI7510 (120 mcg RSV sF plus 5.0 mcg glucopyranosyl lipid A in 2% volume per volume stable emulsion) plus placebo administered by IM injection in contralateral arms on Day 1.
- MEDI7510 (120 mcg sF + 5 mcg GLA)+ IIV, Cohort 3: Participants received single dose of MEDI7510 (120 mcg RSV sF plus 5.0 mcg glucopyranosyl lipid A in 2% volume per volume stable emulsion) plus IIV administered by IM injection in contralateral arms on Day 1.
Period: Overall Study
Arm/Group | MEDI7510 (120 mcg sF + 1 mcg GLA), Cohort 1 | MEDI7510 (80 mcg sF + 2.5 mcg GLA), Cohort 4 | Inactivated Influenza Vaccine (IIV) | MEDI7510 (120 mcg sF + 2.5 mcg GLA) + Placebo, Cohort 2 | MEDI7510 (120 mcg sF + 2.5 mcg GLA) + IIV, Cohort 2 | MEDI7510 (120 mcg sF + 5 mcg GLA) + Placebo, Cohort 3 | MEDI7510 (120 mcg sF + 5 mcg GLA)+ IIV, Cohort 3
Started | 39 | 20 | 44 | 39 | 40 | 40 | 39
Completed | 37 | 18 | 38 | 37 | 40 | 39 | 37
Not Completed | 2 | 2 | 6 | 2 | 0 | 1 | 2
Not completed — Withdrawal by Subject | 2 | 1 | 2 | 1 | 0 | 0 | 1
Not completed — Death | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 3 | 1 | 0 | 1 | 1
Not completed — withdrawal of consent | 0 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MEDI7510 (120 mcg sF + 1 mcg GLA), Cohort 1 | Inactivated Influenza Vaccine (IIV) | MEDI7510 (120 mcg sF + 2.5 mcg GLA) + Placebo, Cohort 2 | MEDI7510 (120 mcg sF + 2.5 mcg GLA) + IIV, Cohort 2 | MEDI7510 (120 mcg sF + 5 mcg GLA) + Placebo, Cohort 3 | MEDI7510 (120 mcg sF + 5 mcg GLA)+ IIV, Cohort 3 | MEDI7510 (80 mcg sF + 2.5 mcg GLA), Cohort 4 | Total
Number analyzed (Participants) | 39 | 44 | 39 | 40 | 40 | 39 | 20 | 261
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.5 (6.9) | 69.6 (7.0) | 69.3 (5.2) | 67.9 (5.8) | 70.1 (5.9) | 70.2 (6.8) | 68.9 (6.5) | 69.5 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 25 | 27 | 19 | 18 | 19 | 13 | 142
  Male | 18 | 19 | 12 | 21 | 22 | 20 | 7 | 119

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Solicited Symptoms
Description: Solicited symptoms are events that are considered likely to occur post dosing and included the local reaction (pain, tenderness or soreness, redness, and swelling at the site of injection) to investigational product (IP) injection and systemic symptoms (fever greater than or equal to [>=] 100.4°F [>=38°C] by any route, headache, generalized muscle aches, and fatigue or tiredness) that might be related to IP injection. Solicited symptoms were not coded using Medical Dictionary for Regulatory Activities (MedDRA) and summarized regardless of whether or not they are treatment emergent. The percentage of participants with solicited symptoms were recorded during Days 1 (day of dosing) through 7.
Time Frame: Day 1 to Day 7
Population: As-treated Population (ATP) included all participants who received any amount of study drug.
Measure: Number; unit: Percentage of Participants
Groups:
- MEDI7510 (120 mcg sF + 5 mcg GLA) + IIV, Cohort 3: Participants received single dose of MEDI7510 (120 mcg RSV sF plus 5.0 mcg glucopyranosyl lipid A in 2% volume per volume stable emulsion) plus IIV administered by IM injection in contralateral arms on Day 1.
Arm/Group | MEDI7510 (120 mcg sF + 1 mcg GLA), Cohort 1 | MEDI7510 (120 mcg sF + 2.5 mcg GLA) + Placebo, Cohort 2 | MEDI7510 (120 mcg sF + 2.5 mcg GLA) + IIV, Cohort 2 | MEDI7510 (80 mcg sF + 2.5 mcg GLA), Cohort 4 | Inactivated Influenza Vaccine (IIV) | MEDI7510 (120 mcg sF + 5 mcg GLA) + Placebo, Cohort 3 | MEDI7510 (120 mcg sF + 5 mcg GLA) + IIV, Cohort 3
Number analyzed (Participants) | 39 | 38 | 40 | 20 | 44 | 40 | 38
Percentage of Participants | 35.9 | 73.7 | 60.0 | 60.0 | 63.6 | 75.0 | 68.4

2. Primary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. Treatment-emergent were the events between administration of study drug and including the follow-up period through Day 29. The AEs were summarized using the Medical Dictionary for Regulatory Activities version 18.1.
Time Frame: From Day 1 to Day 29
Population: ATP included all participants who received any amount of study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | MEDI7510 (120 mcg sF + 1 mcg GLA), Cohort 1 | MEDI7510 (120 mcg sF + 2.5 mcg GLA) + Placebo, Cohort 2 | MEDI7510 (120 mcg sF + 2.5 mcg GLA) + IIV, Cohort 2 | MEDI7510 (80 mcg sF + 2.5 mcg GLA), Cohort 4 | Inactivated Influenza Vaccine (IIV) | MEDI7510 (120 mcg sF + 5 mcg GLA) + Placebo, Cohort 3 | MEDI7510 (120 mcg sF + 5 mcg GLA) + IIV, Cohort 3
Number analyzed (Participants) | 39 | 39 | 40 | 20 | 44 | 40 | 39
Percentage of Participants | 5.1 | 15.4 | 22.5 | 30.0 | 18.2 | 27.5 | 20.5

3. Primary Outcome: Percentage of Participants With Treatment-emergent Serious Adverse Events
Description: A serious adverse event (SAE) was an AE resulting in any of following reason: death, initial or prolonged inpatient hospitalization, life-threatening experience (immediate risk), persistent or significant disability/incapacity, congenital anomaly, and a medical event that may jeopardize the participant or may require medical intervention to prevent one of the outcomes listed above.
Time Frame: From Day 1 to Day 361
Population: ATP included all participants who received any amount of study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | MEDI7510 (120 mcg sF + 1 mcg GLA), Cohort 1 | MEDI7510 (120 mcg sF + 2.5 mcg GLA) + Placebo, Cohort 2 | MEDI7510 (120 mcg sF + 2.5 mcg GLA) + IIV, Cohort 2 | MEDI7510 (80 mcg sF + 2.5 mcg GLA), Cohort 4 | Inactivated Influenza Vaccine (IIV) | MEDI7510 (120 mcg sF + 5 mcg GLA) + Placebo, Cohort 3 | MEDI7510 (120 mcg sF + 5 mcg GLA) + IIV, Cohort 3
Number analyzed (Participants) | 39 | 39 | 40 | 20 | 44 | 40 | 39
Percentage of Participants | 2.6 | 5.1 | 0 | 0 | 2.3 | 0 | 2.6

4. Primary Outcome: Percentage of Participants With New Onset Chronic Diseases (NOCDs)
Description: A NOCD was a newly diagnosed medical condition that is of a chronic, ongoing nature. It was observed after receiving study drug and was assessed by investigator as medically significant. All NOCDs were recorded from the time of dosing through the day of the last participant contact (Day 361 visit).
Time Frame: From Day 1 to Day 361
Population: ATP included all participants who received any amount of study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | MEDI7510 (120 mcg sF + 1 mcg GLA), Cohort 1 | MEDI7510 (120 mcg sF + 2.5 mcg GLA) + Placebo, Cohort 2 | MEDI7510 (120 mcg sF + 2.5 mcg GLA) + IIV, Cohort 2 | MEDI7510 (80 mcg sF + 2.5 mcg GLA), Cohort 4 | Inactivated Influenza Vaccine (IIV) | MEDI7510 (120 mcg sF + 5 mcg GLA) + Placebo, Cohort 3 | MEDI7510 (120 mcg sF + 5 mcg GLA) + IIV, Cohort 3
Number analyzed (Participants) | 39 | 39 | 40 | 20 | 44 | 40 | 39
Percentage of Participants | 2.6 | 0 | 5.0 | 5.0 | 0 | 0 | 0

5. Primary Outcome: Percentage of Participants With Treatment-emergent Adverse Events of Special Interest (TEAESI)
Description: An AESI was one of scientific and medical interest specific to understanding of study product and may have required close monitoring and rapid communication by investigator to the sponsor. Treatment emergent AESIs were collected from the time of dosing through the day of the last participant contact (Day 361 visit).
Time Frame: From Day 1 to Day 361
Population: ATP included all participants who received any amount of study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | MEDI7510 (120 mcg sF + 1 mcg GLA), Cohort 1 | MEDI7510 (120 mcg sF + 2.5 mcg GLA) + Placebo, Cohort 2 | MEDI7510 (120 mcg sF + 2.5 mcg GLA) + IIV, Cohort 2 | MEDI7510 (80 mcg sF + 2.5 mcg GLA), Cohort 4 | Inactivated Influenza Vaccine (IIV) | MEDI7510 (120 mcg sF + 5 mcg GLA) + Placebo, Cohort 3 | MEDI7510 (120 mcg sF + 5 mcg GLA) + IIV, Cohort 3
Number analyzed (Participants) | 39 | 39 | 40 | 20 | 44 | 40 | 39
Percentage of Participants | 0 | 0 | 0 | 0 | 0 | 2.5 | 0

6. Secondary Outcome: Geometric Mean Titers (GMTs) of Serum Antibodies Against Respiratory Syncytial Virus (RSV) by RSV A Microneutralization Assay
Description: GMTs of serum antibodies against RSV, as assessed by the RSV A microneutralization assay at Baseline and the results through Day 361 were presented. Humoral immunogenicity samples was used to assess RSV A neutralizing antibody. Humoral immunity against RSV was assessed by a microneutralization assay for RSV A. Immunogenicity population is defined as all participants in ATP who had no protocol deviation judged to have the potential to interfere with generation or interpretation of an immune response.
Time Frame: Baseline (Day 1), Day 29, 61, 91, 181, 271, and 361
Population: Immunogenicity population
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | MEDI7510 (120 mcg sF + 1 mcg GLA), Cohort 1 | MEDI7510 (120 mcg sF + 2.5 mcg GLA) + Placebo, Cohort 2 | MEDI7510 (120 mcg sF + 2.5 mcg GLA) + IIV, Cohort 2 | MEDI7510 (80 mcg sF + 2.5 mcg GLA), Cohort 4 | Inactivated Influenza Vaccine (IIV) | MEDI7510 (120 mcg sF + 5 mcg GLA) + Placebo, Cohort 3 | MEDI7510 (120 mcg sF + 5 mcg GLA) + IIV, Cohort 3
Number analyzed (Participants) | 39 | 39 | 40 | 20 | 44 | 40 | 38
Titers
  Baseline (Day 1) | 441.15 [344.99 to 564.11] | 397.52 [279.60 to 565.17] | 401.85 [313.66 to 514.82] | 504.78 [332.66 to 765.95] | 513.53 [414.42 to 636.36] | 365.19 [275.62 to 483.87] | 510.88 [416.00 to 627.40]
  Day 29: number analyzed (Participants) | 39 | 38 | 40 | 20 | 43 | 40 | 37
  Day 29 | 1068.43 [820.93 to 1390.57] | 1233.62 [1010.37 to 1506.21] | 1004.49 [839.19 to 1202.36] | 1217.75 [867.21 to 1709.98] | 464.13 [372.16 to 578.82] | 958.74 [792.78 to 1159.45] | 1370.55 [1115.61 to 1683.75]
  Day 61: number analyzed (Participants) | 39 | 0 | 0 | 20 | 43 | 40 | 36
  Day 61 | 1168.56 [915.50 to 1491.57] |  |  | 1081.64 [750.47 to 1558.93] | 626.09 [509.37 to 769.57] | 816.33 [676.78 to 984.64] | 1151.62 [939.64 to 1411.41]
  Day 91: number analyzed (Participants) | 39 | 0 | 0 | 20 | 42 | 40 | 37
  Day 91 | 1078.35 [839.60 to 1385.00] |  |  | 967.42 [665.58 to 1406.14] | 579.56 [463.07 to 725.34] | 765.63 [642.61 to 912.20] | 1072.70 [854.84 to 1346.08]
  Day 181: number analyzed (Participants) | 36 | 0 | 0 | 20 | 40 | 40 | 36
  Day 181 | 866.23 [673.55 to 1114.04] |  |  | 763.51 [514.29 to 1133.49] | 548.46 [439.44 to 684.53] | 631.44 [511.84 to 778.99] | 900.59 [716.04 to 1132.70]
  Day 271: number analyzed (Participants) | 36 | 0 | 0 | 19 | 39 | 39 | 33
  Day 271 | 796.48 [607.83 to 1043.70] |  |  | 579.19 [329.21 to 1018.98] | 546.80 [435.46 to 686.62] | 565.08 [460.42 to 693.53] | 690.36 [552.52 to 862.59]
  Day 361: number analyzed (Participants) | 36 | 0 | 0 | 18 | 34 | 38 | 35
  Day 361 | 746.01 [594.45 to 936.22] |  |  | 814.32 [515.32 to 1286.80] | 573.22 [458.58 to 716.51] | 533.55 [426.01 to 668.23] | 692.93 [554.05 to 866.62]

7. Secondary Outcome: Geometric Mean Fold Rises (GMFRs) of Serum Antibodies Against RSV by RSV A Microneutralization Assay
Description: GMFRs of serum antibodies against RSV, as assessed by the RSV A microneutralization assay from Baseline line through Day 361 were presented. Humoral immunogenicity samples was used to assess RSV A neutralizing antibody. Humoral immunity against RSV was assessed by a microneutralization assay for RSV A.
Time Frame: Day 29, 61, 91, 181, 271, and 361
Population: Immunogenicity Population. Here, 'n' is number of participants analyzed for this outcome measure at given time points.
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | MEDI7510 (120 mcg sF + 1 mcg GLA), Cohort 1 | MEDI7510 (120 mcg sF + 2.5 mcg GLA) + Placebo, Cohort 2 | MEDI7510 (120 mcg sF + 2.5 mcg GLA) + IIV, Cohort 2 | MEDI7510 (80 mcg sF + 2.5 mcg GLA), Cohort 4 | Inactivated Influenza Vaccine (IIV) | MEDI7510 (120 mcg sF + 5 mcg GLA) + Placebo, Cohort 3 | MEDI7510 (120 mcg sF + 5 mcg GLA) + IIV, Cohort 3
Number analyzed (Participants) | 39 | 39 | 40 | 20 | 44 | 40 | 38
Fold rise
  Day 29: number analyzed (Participants) | 39 | 38 | 40 | 20 | 43 | 40 | 37
  Day 29 | 2.42 [1.96 to 2.99] | 3.26 [2.29 to 4.63] | 2.50 [2.11 to 2.97] | 2.41 [1.82 to 3.20] | 0.92 [0.86 to 0.97] | 2.63 [2.17 to 3.18] | 2.64 [2.12 to 3.30]
  Day 61: number analyzed (Participants) | 39 | 0 | 0 | 20 | 43 | 40 | 36
  Day 61 | 2.65 [2.21 to 3.17] |  |  | 2.14 [1.60 to 2.87] | 1.24 [1.08 to 1.42] | 2.24 [1.81 to 2.76] | 2.20 [1.79 to 2.70]
  Day 91: number analyzed (Participants) | 39 | 0 | 0 | 20 | 42 | 40 | 37
  Day 91 | 2.44 [2.05 to 2.92] |  |  | 1.92 [1.43 to 2.56] | 1.14 [1.04 to 1.25] | 2.10 [1.70 to 2.59] | 2.07 [1.65 to 2.59]
  Day 181: number analyzed (Participants) | 36 | 0 | 0 | 20 | 40 | 40 | 36
  Day 181 | 1.99 [1.72 to 2.30] |  |  | 1.51 [1.20 to 1.91] | 1.15 [1.02 to 1.30] | 1.73 [1.44 to 2.08] | 1.68 [1.37 to 2.06]
  Day 271: number analyzed (Participants) | 36 | 0 | 0 | 19 | 39 | 39 | 33
  Day 271 | 1.83 [1.57 to 2.14] |  |  | 1.08 [0.64 to 1.81] | 1.11 [0.96 to 1.27] | 1.56 [1.32 to 1.86] | 1.42 [1.18 to 1.70]
  Day 361: number analyzed (Participants) | 36 | 0 | 0 | 18 | 34 | 38 | 35
  Day 361 | 1.71 [1.50 to 1.96] |  |  | 1.47 [1.12 to 1.93] | 1.15 [1.00 to 1.31] | 1.50 [1.27 to 1.77] | 1.34 [1.14 to 1.56]

8. Secondary Outcome: Percentage of Participants With Post-dose Seroresponse to RSV by RSV A Microneutralization Assay
Description: Seroresponse defined as a greater than or equal to (>=) 3-fold rise in titer from baseline. Humoral immunogenicity samples was used to assess RSV A neutralizing antibody. Humoral immunity against RSV was assessed by a microneutralization assay for RSV A.
Time Frame: Day 29
Population: Immunogenicity population.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | MEDI7510 (120 mcg sF + 1 mcg GLA), Cohort 1 | MEDI7510 (120 mcg sF + 2.5 mcg GLA) + Placebo, Cohort 2 | MEDI7510 (120 mcg sF + 2.5 mcg GLA) + IIV, Cohort 2 | MEDI7510 (80 mcg sF + 2.5 mcg GLA), Cohort 4 | Inactivated Influenza Vaccine (IIV) | MEDI7510 (120 mcg sF + 5 mcg GLA) + Placebo, Cohort 3 | MEDI7510 (120 mcg sF + 5 mcg GLA) + IIV, Cohort 3
Number analyzed (Participants) | 39 | 39 | 40 | 20 | 44 | 40 | 38
Percentage of Participants | 41.0 [25.57 to 57.90] | 42.1 [26.31 to 59.18] | 42.5 [27.04 to 59.11] | 30.0 [11.89 to 54.28] | 0 [0.00 to 8.22] | 35.0 [20.63 to 51.68] | 40.5 [24.75 to 57.90]

9. Secondary Outcome: Geometric Mean Concentrations of Serum Antibodies Against RSV by Anti F Immunoglobulin G (IgG) Assay
Description: Humoral immunogenicity samples were used to assess anti-F IgG antibodies measured using a 4-plex Meso Scale Discovery (MSD) platform assay. Results through Day 361 are presented.
Time Frame: Baseline (Day 1), Day 29, 61, 91, 181, 271, and 361
Population: Immunogenicity Population. Here, 'n' is number of participants analyzed for this outcome measure at given time points.
Measure: Geometric Mean (95% Confidence Interval); unit: F Ab Unit/mL
Arm/Group | MEDI7510 (120 mcg sF + 1 mcg GLA), Cohort 1 | MEDI7510 (120 mcg sF + 2.5 mcg GLA) + Placebo, Cohort 2 | MEDI7510 (120 mcg sF + 2.5 mcg GLA) + IIV, Cohort 2 | MEDI7510 (80 mcg sF + 2.5 mcg GLA), Cohort 4 | Inactivated Influenza Vaccine (IIV) | MEDI7510 (120 mcg sF + 5 mcg GLA) + Placebo, Cohort 3 | MEDI7510 (120 mcg sF + 5 mcg GLA) + IIV, Cohort 3
Number analyzed (Participants) | 39 | 39 | 40 | 20 | 44 | 40 | 38
F Ab Unit/mL
  Baseline (Day 1) | 99.63 [74.22 to 133.73] | 95.29 [62.83 to 144.54] | 101.51 [75.45 to 136.58] | 67.93 [30.62 to 150.71] | 92.34 [76.64 to 111.25] | 70.18 [55.27 to 89.11] | 82.13 [64.16 to 105.14]
  Day 29: number analyzed (Participants) | 39 | 38 | 40 | 20 | 43 | 40 | 37
  Day 29 | 1328.36 [958.76 to 1840.45] | 1433.98 [1053.24 to 1952.34] | 1047.68 [810.79 to 1353.79] | 1003.07 [566.77 to 1775.23] | 92.94 [76.81 to 112.46] | 1066.90 [836.10 to 1361.42] | 1474.47 [1110.41 to 1957.90]
  Day 61: number analyzed (Participants) | 39 | 0 | 0 | 20 | 42 | 40 | 37
  Day 61 | 1050.29 [774.32 to 1424.61] |  |  | 852.27 [491.53 to 1477.76] | 104.00 [80.54 to 134.30] | 850.91 [661.84 to 1093.99] | 1097.04 [816.40 to 1474.15]
  Day 91: number analyzed (Participants) | 39 | 0 | 0 | 20 | 41 | 40 | 37
  Day 91 | 817.05 [603.67 to 1105.86] |  |  | 662.15 [375.50 to 1167.62] | 95.29 [77.73 to 116.82] | 705.96 [547.07 to 910.99] | 845.04 [636.42 to 1122.04]
  Day 181: number analyzed (Participants) | 36 | 0 | 0 | 20 | 40 | 40 | 36
  Day 181 | 501.47 [368.62 to 682.20] |  |  | 403.58 [226.56 to 718.92] | 91.54 [74.62 to 112.29] | 466.81 [363.97 to 598.71] | 531.43 [398.10 to 709.41]
  Day 271: number analyzed (Participants) | 36 | 0 | 0 | 19 | 39 | 39 | 33
  Day 271 | 389.94 [286.92 to 529.96] |  |  | 341.99 [160.13 to 730.40] | 92.70 [75.46 to 113.88] | 356.11 [276.99 to 457.84] | 423.30 [316.79 to 565.61]
  Day 361: number analyzed (Participants) | 36 | 0 | 0 | 18 | 34 | 38 | 35
  Day 361 | 343.64 [255.99 to 461.32] |  |  | 284.56 [140.69 to 575.55] | 94.10 [74.03 to 119.61] | 305.10 [235.90 to 394.60] | 354.13 [268.29 to 467.43]

10. Secondary Outcome: GMFRs of Serum Antibodies Against RSV by Anti F IgG Assay
Description: The Anti F IgG antibodies were derived from the RSV-specific 4-plex MSD assay developed on the Meso Scale discovery platform. Humoral immunogenicity samples were used to assess anti-F IgG antibodies measured using a 4-plex Meso Scale Discovery (MSD) platform assay. Results through Day 361 are presented.
Time Frame: Day 29, 61, 91, 181, 271, and 361
Population: Immunogenicity Population. Here, 'n' is number of participants analyzed for this outcome measure at given time points.
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | MEDI7510 (120 mcg sF + 1 mcg GLA), Cohort 1 | MEDI7510 (120 mcg sF + 2.5 mcg GLA) + Placebo, Cohort 2 | MEDI7510 (120 mcg sF + 2.5 mcg GLA) + IIV, Cohort 2 | MEDI7510 (80 mcg sF + 2.5 mcg GLA), Cohort 4 | Inactivated Influenza Vaccine (IIV) | MEDI7510 (120 mcg sF + 5 mcg GLA) + Placebo, Cohort 3 | MEDI7510 (120 mcg sF + 5 mcg GLA) + IIV, Cohort 3
Number analyzed (Participants) | 39 | 39 | 40 | 20 | 44 | 40 | 38
Fold rise
  Day 29: number analyzed (Participants) | 39 | 38 | 40 | 20 | 43 | 40 | 37
  Day 29 | 13.33 [9.39 to 18.93] | 15.15 [10.18 to 22.55] | 10.32 [7.87 to 13.54] | 14.77 [7.63 to 28.59] | 0.99 [0.96 to 1.02] | 15.20 [11.29 to 20.47] | 17.95 [14.06 to 22.91]
  Day 61: number analyzed (Participants) | 39 | 0 | 0 | 20 | 42 | 40 | 37
  Day 61 | 10.54 [7.73 to 14.37] |  |  | 12.55 [6.55 to 24.04] | 1.09 [0.91 to 1.32] | 12.13 [9.20 to 15.98] | 13.35 [10.51 to 16.96]
  Day 91: number analyzed (Participants) | 39 | 0 | 0 | 20 | 41 | 40 | 37
  Day 91 | 8.20 [6.09 to 11.05] |  |  | 9.75 [5.37 to 17.70] | 1.00 [0.95 to 1.05] | 10.06 [7.74 to 13.07] | 10.28 [8.18 to 12.94]
  Day 181: number analyzed (Participants) | 36 | 0 | 0 | 20 | 40 | 40 | 36
  Day 181 | 5.03 [3.89 to 6.50] |  |  | 5.94 [3.58 to 9.85] | 0.97 [0.92 to 1.02] | 6.65 [5.23 to 8.47] | 6.23 [5.01 to 7.74]
  Day 271: number analyzed (Participants) | 36 | 0 | 0 | 19 | 39 | 39 | 33
  Day 271 | 3.91 [3.05 to 5.02] |  |  | 4.92 [3.11 to 7.77] | 0.96 [0.91 to 1.01] | 5.14 [4.09 to 6.44] | 4.75 [3.76 to 5.99]
  Day 361: number analyzed (Participants) | 36 | 0 | 0 | 18 | 34 | 38 | 35
  Day 361 | 3.45 [2.74 to 4.33] |  |  | 4.22 [2.61 to 6.80] | 0.96 [0.91 to 1.02] | 4.47 [3.55 to 5.65] | 4.07 [3.29 to 5.03]

11. Secondary Outcome: Percentage of Participants With Post-dose Seroresponse to RSV by Anti-F IgG Assay
Description: Seroresponse defined as a greater than or equal to (>=) 3-fold rise from baseline. Humoral immunity against RSV was assessed by an Anti-F IgG assay derived from the RSV-specific 4-plex MSD assay.
Time Frame: Day 29
Population: Immunogenicity population.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | MEDI7510 (120 mcg sF + 1 mcg GLA), Cohort 1 | MEDI7510 (120 mcg sF + 2.5 mcg GLA) + Placebo, Cohort 2 | MEDI7510 (120 mcg sF + 2.5 mcg GLA) + IIV, Cohort 2 | MEDI7510 (80 mcg sF + 2.5 mcg GLA), Cohort 4 | Inactivated Influenza Vaccine (IIV) | MEDI7510 (120 mcg sF + 5 mcg GLA) + Placebo, Cohort 3 | MEDI7510 (120 mcg sF + 5 mcg GLA) + IIV, Cohort 3
Number analyzed (Participants) | 39 | 39 | 40 | 20 | 44 | 40 | 38
Percentage of Participants | 94.9 [82.68 to 99.37] | 89.5 [75.20 to 97.06] | 90.0 [76.34 to 97.21] | 85.0 [62.11 to 96.79] | 0 [0.00 to 8.22] | 97.5 [86.84 to 99.94] | 97.3 [85.84 to 99.93]

12. Secondary Outcome: Ratios of GMTs and GMFRs of Hemagglutination Inhibition (HAI) Antibodies
Description: The ratio of post-dose HAI antibody GMTs and GMFRs in the IIV group and the MEDI7510 plus IIV group was provided by strain and by cohort for Cohorts 2 and 3 to check the effect of MEDI7510 on IIV when administered together. Humoral immunity against influenza consisting of HAI antibody to strains antigenically matched to those contained in the IIV was assessed on Day 29 by each strain (H1N1, H3N2, B/Yamagata).
Time Frame: Day 29
Population: Immunogenicity Population.
Measure: Number (95% Confidence Interval); unit: Ratio
Arm/Group | MEDI7510 (120 mcg sF + 2.5 mcg GLA) + Placebo, Cohort 2 | MEDI7510 (120 mcg sF + 2.5 mcg GLA) + IIV, Cohort 2 | MEDI7510 (120 mcg sF + 5 mcg GLA) + Placebo, Cohort 3 | MEDI7510 (120 mcg sF + 5 mcg GLA) + IIV, Cohort 3
Number analyzed (Participants) | 38 | 40 | 40 | 37
Ratio
  GMT: H1N1 | NA [NA to NA] — Data is not available for this time point because the humoral immunity against influenza consisting of HAI antibody to strains antigenically matched to those contained in the IIV was assessed. | 1.19 [0.71 to 1.99] | NA [NA to NA] — Data is not available for this time point because the humoral immunity against influenza consisting of HAI antibody to strains antigenically matched to those contained in the IIV was assessed. | 1.01 [0.63 to 1.61]
  GMT: H3N2 | NA [NA to NA] — Data is not available for this time point because the humoral immunity against influenza consisting of HAI antibody to strains antigenically matched to those contained in the IIV was assessed. | 1.53 [1.03 to 2.28] | NA [NA to NA] — Data is not available for this time point because the humoral immunity against influenza consisting of HAI antibody to strains antigenically matched to those contained in the IIV was assessed. | 0.78 [0.53 to 1.15]
  GMT: B/Yamagata | NA [NA to NA] — Data is not available for this time point because the humoral immunity against influenza consisting of HAI antibody to strains antigenically matched to those contained in the IIV was assessed. | 1.38 [0.81 to 2.36] | NA [NA to NA] — Data is not available for this time point because the humoral immunity against influenza consisting of HAI antibody to strains antigenically matched to those contained in the IIV was assessed. | 1.49 [0.91 to 2.46]
  GMFR: H1N1 | NA [NA to NA] — Data is not available for this time point because the humoral immunity against influenza consisting of HAI antibody to strains antigenically matched to those contained in the IIV was assessed. | 1.13 [0.68 to 1.87] | NA [NA to NA] — Data is not available for this time point because the humoral immunity against influenza consisting of HAI antibody to strains antigenically matched to those contained in the IIV was assessed. | 0.97 [0.54 to 1.75]
  GMFR: H3N2 | NA [NA to NA] — Data is not available for this time point because the humoral immunity against influenza consisting of HAI antibody to strains antigenically matched to those contained in the IIV was assessed. | 1.53 [0.86 to 2.72] | NA [NA to NA] — Data is not available for this time point because the humoral immunity against influenza consisting of HAI antibody to strains antigenically matched to those contained in the IIV was assessed. | 1.28 [0.69 to 2.38]
  GMFR: B/Yamagata | NA [NA to NA] — Data is not available for this time point because the humoral immunity against influenza consisting of HAI antibody to strains antigenically matched to those contained in the IIV was assessed. | 1.09 [0.76 to 1.55] | NA [NA to NA] — Data is not available for this time point because the humoral immunity against influenza consisting of HAI antibody to strains antigenically matched to those contained in the IIV was assessed. | 1.00 [0.71 to 1.40]

13. Secondary Outcome: Geometric Mean Counts of Cellular Immune Response Against RSV by Respiratory Syncytial Virus Fusion Protein (RSV F) Interferon Gamma (IFNγ) Enzyme-linked Immunosorbent Spot (ELISPOT) Assay
Description: The Geometric Mean Counts assessed by the ELISPOT assay for F protein-specific gamma interferon-producing T cells was performed using RSV F peptides. Cell-mediated immunity was assessed using an IFNγ ELISPOT assay to measure the T-cell responses to the RSV F peptide pool using thawed, cryopreserved peripheral blood mononuclear cell samples.
Time Frame: Baseline (Day 1) and Day 8
Population: Immunogenicity Population. Here, 'n' is number of participants analyzed for this outcome measure at given time points.
Measure: Geometric Mean (95% Confidence Interval); unit: Spot forming counts per 10^6 PBMCs
Arm/Group | MEDI7510 (120 mcg sF + 1 mcg GLA), Cohort 1 | MEDI7510 (120 mcg sF + 2.5 mcg GLA) + Placebo, Cohort 2 | MEDI7510 (120 mcg sF + 2.5 mcg GLA) + IIV, Cohort 2 | MEDI7510 (80 mcg sF + 2.5 mcg GLA), Cohort 4 | Inactivated Influenza Vaccine (IIV) | MEDI7510 (120 mcg sF + 5 mcg GLA) + Placebo, Cohort 3 | MEDI7510 (120 mcg sF + 5 mcg GLA) + IIV, Cohort 3
Number analyzed (Participants) | 38 | 37 | 34 | 20 | 39 | 40 | 38
Spot forming counts per 10^6 PBMCs
  Baseline (Day 1): number analyzed (Participants) | 34 | 32 | 33 | 20 | 36 | 40 | 36
  Baseline (Day 1) | 66.06 [53.40 to 81.72] | 47.21 [39.96 to 55.77] | 50.89 [42.19 to 61.38] | 42.24 [33.84 to 52.73] | 58.53 [47.10 to 72.74] | 45.71 [38.90 to 53.71] | 62.63 [49.89 to 78.61]
  Day 8: number analyzed (Participants) | 38 | 31 | 31 | 19 | 35 | 40 | 36
  Day 8 | 436.72 [333.87 to 571.25] | 341.02 [222.54 to 522.58] | 430.33 [308.22 to 600.83] | 379.28 [225.90 to 636.80] | 54.30 [43.86 to 67.24] | 376.43 [273.42 to 518.25] | 618.15 [463.46 to 824.48]

14. Secondary Outcome: GMFRs of Cellular Immune Response Against RSV by RSV F IFNγ ELISPOT Assay
Description: The GMFRs assessed by the ELISPOT assay for F protein-specific gamma interferon-producing T cells was performed using RSV F peptides. Cell-mediated immunity was assessed using an IFNγ ELISPOT assay to measure the T-cell responses to the RSV F peptide pool using thawed, cryopreserved peripheral blood mononuclear cell samples
Time Frame: Day 8
Population: Immunogenicity Population.
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | MEDI7510 (120 mcg sF + 1 mcg GLA), Cohort 1 | MEDI7510 (120 mcg sF + 2.5 mcg GLA) + Placebo, Cohort 2 | MEDI7510 (120 mcg sF + 2.5 mcg GLA) + IIV, Cohort 2 | MEDI7510 (80 mcg sF + 2.5 mcg GLA), Cohort 4 | Inactivated Influenza Vaccine (IIV) | MEDI7510 (120 mcg sF + 5 mcg GLA) + Placebo, Cohort 3 | MEDI7510 (120 mcg sF + 5 mcg GLA) + IIV, Cohort 3
Number analyzed (Participants) | 34 | 26 | 30 | 19 | 32 | 40 | 35
Fold rise | 6.45 [4.88 to 8.52] | 6.77 [4.13 to 11.09] | 8.67 [6.38 to 11.78] | 8.87 [4.99 to 15.77] | 0.89 [0.76 to 1.04] | 8.23 [5.92 to 11.46] | 10.48 [7.82 to 14.03]

15. Secondary Outcome: Percentage of Participants With Post-dose Cell-mediated Immune Response to RSV F by RSV F Peptide Pool IFNγ ELISPOT
Description: Seroresponse defined as a greater than or equal to (>=) 3-fold rise from baseline. The Cell-mediated immunity was assessed using an IFNγ ELISPOT assay to measure the T-cell responses to the RSV F peptide pool using thawed, cryopreserved peripheral blood mononuclear cell samples.
Time Frame: Day 8
Population: Immunogenicity Population.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | MEDI7510 (120 mcg sF + 1 mcg GLA), Cohort 1 | MEDI7510 (120 mcg sF + 2.5 mcg GLA) + Placebo, Cohort 2 | MEDI7510 (120 mcg sF + 2.5 mcg GLA) + IIV, Cohort 2 | MEDI7510 (80 mcg sF + 2.5 mcg GLA), Cohort 4 | Inactivated Influenza Vaccine (IIV) | MEDI7510 (120 mcg sF + 5 mcg GLA) + Placebo, Cohort 3 | MEDI7510 (120 mcg sF + 5 mcg GLA) + IIV, Cohort 3
Number analyzed (Participants) | 34 | 26 | 30 | 19 | 32 | 40 | 35
Percentage of Participants | 76.5 [58.83 to 89.25] | 80.8 [60.65 to 93.45] | 90.0 [73.47 to 97.89] | 78.9 [54.43 to 93.95] | 0.00 [0.00 to 10.89] | 82.5 [67.22 to 92.66] | 97.1 [85.08 to 99.93]

ADVERSE EVENTS:
Time Frame: AEs and SAEs were collected from time of signature of informed consent throughout the treatment period and including the follow-up period through the Day 29 visit and day of last subject contact (Day 361 visit), respectively
Arm/Group | MEDI7510 (120 mcg sF + 1 mcg GLA), Cohort 1 | Inactivated Influenza Vaccine (IIV) | MEDI7510 (120 mcg sF + 2.5 mcg GLA) + Placebo, Cohort 2 | MEDI7510 (120 mcg sF + 2.5 mcg GLA) + IIV, Cohort 2 | MEDI7510 (120 mcg sF + 5 mcg GLA) + Placebo, Cohort 3 | MEDI7510 (120 mcg sF + 5 mcg GLA)+ IIV, Cohort 3 | MEDI7510 (80 mcg sF + 2.5 mcg GLA), Cohort 4
Serious Adverse Events (participants affected / at risk) | 1/39 | 1/44 | 2/39 | 0/40 | 0/40 | 1/39 | 0/20
Other Adverse Events (participants affected / at risk) | 2/39 | 8/44 | 5/39 | 9/40 | 11/40 | 8/39 | 6/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MEDI7510 (120 mcg sF + 1 mcg GLA), Cohort 1 (N=39) | Inactivated Influenza Vaccine (IIV) (N=44) | MEDI7510 (120 mcg sF + 2.5 mcg GLA) + Placebo, Cohort 2 (N=39) | MEDI7510 (120 mcg sF + 2.5 mcg GLA) + IIV, Cohort 2 (N=40) | MEDI7510 (120 mcg sF + 5 mcg GLA) + Placebo, Cohort 3 (N=40) | MEDI7510 (120 mcg sF + 5 mcg GLA)+ IIV, Cohort 3 (N=39) | MEDI7510 (80 mcg sF + 2.5 mcg GLA), Cohort 4 (N=20)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MEDI7510 (120 mcg sF + 1 mcg GLA), Cohort 1 (N=39) | Inactivated Influenza Vaccine (IIV) (N=44) | MEDI7510 (120 mcg sF + 2.5 mcg GLA) + Placebo, Cohort 2 (N=39) | MEDI7510 (120 mcg sF + 2.5 mcg GLA) + IIV, Cohort 2 (N=40) | MEDI7510 (120 mcg sF + 5 mcg GLA) + Placebo, Cohort 3 (N=40) | MEDI7510 (120 mcg sF + 5 mcg GLA)+ IIV, Cohort 3 (N=39) | MEDI7510 (80 mcg sF + 2.5 mcg GLA), Cohort 4 (N=20)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blepharospasm (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Iridocyclitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Axillary pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bone contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Wound haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary hesitation (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.